CLINICAL TRIAL: NCT03739320
Title: A Prospective Observational Study on the Effect of Mepolizumab add-on Therapy on Daily Physical Activity in Patients With Severe Eosinophilic Asthma
Brief Title: A Study on the Effect of Mepolizumab Therapy on Daily Physical Activity of Patients With Severe Eosinophilic Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sotiria General Hospital (Other)
Responsible Party: Principal Investigator, Marios Panagiotou, Respiratory Physician, PhD student, Sotiria General Hospital
Other Study IDs: 451
Record Dates: First submitted 2018-11-07; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Severe Eosinophilic Asthma
Keywords: severe asthma; biologic therapy; physical activity monitoring
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma | interventions — mepolizumab; Injections

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Mepolizumab 100 MG Injection [Nucala] — 100 milligrams subcutaneously once every 4 weeks

SUMMARY:
Daily physical activity in adult patients with asthma remains overlooked. Limited evidence demonstrates reduced levels of daily physical activity in asthma populations but studies examining the potential effect of available therapies are missing. This study aims to investigate the overall levels of daily physical activity in patients with severe eosinophilic asthma and whether anti-interleukin-5 therapy with mepolizumab, on top of existing, maximal, and optimised asthma treatment, may improve patient's daily physical activity.

DETAILED DESCRIPTION:
A multi-centre, prospective, observational study of continuous patients who fulfil the definition of severe asthma and the criteria for mepolizumab (nucala; GSK) therapy. Patients have their daily physical activity recorded using triaxial accelerometry (DynaPort MoveMonitor; McRoberts) prior to treatment, and at 6 and 12 months of mepolizumab therapy (100 mg subcutaneously once every 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Severe asthma
2. Criteria for mepolizumab therapy: blood eosinophils ≥150 cells/μL at screening or ≥300 cells/μL in the past 12 months.

Exclusion Criteria: Comorbidities limiting physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with severe asthma, already on maximal and optimised treatment who fulfil the criteria for mepolizumab add-on therapy.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in daily moving time | 7 days
  Moving time in minutes
Change in daily movement intensity | 7 days
  Movement intensity in m/s^2
Change in daily time in moderate-to-vigorous-intensity activity | 7 days
  Time in moderate-to-vigorous-intensity activity in minutes
Change in daily steps | 7 days
  Step count

CONTACTS AND LOCATIONS:
Overall Officials: Marios Panagiotou, MD, Principal Investigator — Sotiria General Hospital
Locations (1):
- Sotiria General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided